CLINICAL TRIAL: NCT01548326
Title: Effects of Short-term Atorvastatin Treatment on Vaccination Efficacy in Nonresponder Persons to Hepatitis B Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nematollah Jonaidi Jafari (Other)
Responsible Party: Sponsor-Investigator, Nematollah Jonaidi Jafari, Head of Health Research Center, Baqiyatallah Medical Sciences University
Organization: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: behdasht-90-6-16; IRCT201109147556N1 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Hepatitis B; Vaccination Failure
Keywords: Vaccination Failure; Nonresponder; Hepatitis B virus; Atorvastatin; Immunization against viral Hepatitis
MeSH Terms: conditions — Hepatitis B | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): will receive one 40 mg Atorvastatin tablet orally per day for 10 days and in 5th day 1 dose of recombinant yeast-derived Hepatitis B vaccine intramuscular in left Deltoid muscle
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): will receive one Placebo tablet orally per day for 10 days and in 5th day 1 dose of recombinant yeast-derived Hepatitis B vaccine intramuscular in left Deltoid muscle
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atorvastatin — one 40 mg Atorvastatin tablet orally per day for 10 days
  Arms: Atorvastatin
Drug: placebo — one Placebo tablet orally per day for 10 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether short-term Atorvastatin can increase the immunity response to hepatitis B vaccination in vaccine Nonresponders.

DETAILED DESCRIPTION:
20 person of vaccinated individuals who have HBsAb<10 after 3 dose hepatitis B vaccination who called Nonresponders will be randomly allocated in 2 groups. one group receive short-term Atorvastatin and other group receive placebo.both group will be vaccinated with hepatitis B vaccine and then immunity response will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Previous 3 dose hepatitis B vaccination
* Negative HBc Ab
* Negative HBs Ag
* HBs Ab less than 10 in ELIZA

Exclusion Criteria:

* positive serologic evidence of Hepatitis B infection
* Chronic use of Atorvastatin
* Immunosuppressive Disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum HBsAb level | 1 month after vaccination
  HBsAb level in serum measurement with quantitative ELIZA method

SECONDARY OUTCOMES:
IL-4 level in WBC culture | 1 month after vaccination
  IL-4 level measurement with polymerase chain reaction method
IL 17 level in WBC culture | 1 month after vaccination
  IL 17 level measurement with polymerase chain reaction method
TGF-beta level in WBC culture | 1 month after vaccination
  TGF-beta level measurement with polymerase chain reaction method
IFN-gamma level in WBC culture | 1 month after vaccination
  IFN-gamma level measurement with polymerase chain reaction method

CONTACTS AND LOCATIONS:
Overall Officials: Nematollah Jonaidi Jafari, MD, Study Chair — Baqiyatallah University of Medical Sciencesc
Locations (1):
- Baqiyatallah University of Medical Sciences, Tehran, Tehran Province, Iran